CLINICAL TRIAL: NCT04451681
Title: Evaluation of Physical Performance in Ankylosing Spondylitis Patients by Cardiopulmonary Exercise Test
Brief Title: Evaluation of Physical Performance in Ankylosing Spondylitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BVUFTRAS1
Record Dates: First submitted 2020-06-19; First posted 2020-06-30 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing spondylitis; Cardiopulmonary exercise test; Aerobic physical capacity; VO2max
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankylosing spondylitis (Other): A total of 42 patients, who were diagnosed with AS with modified New York Criteria, and who agreed to participate in the study, will be included in this group.
  Interventions: Other: Cardiopulmonary exercise test
- Control (Other): A total of 42 control participants between the ages of 18-65 who agreed to participate in the study will be included in this group.
  Interventions: Other: Cardiopulmonary exercise test

INTERVENTIONS:
Other: Cardiopulmonary exercise test — Data such as oxygen consumption, cardiac parameters and speed of the patient are analyzed numerically on the treadmill in the KPET; Objective performance values such as maximum oxygen use (VO2max), maximum heart rate, respiratory capacity, and maximum rate will be obtained.

SUMMARY:
Ankylosing spondylitis (AS) can cause serious limitations in individuals' physical performance, as it involves the musculoskeletal system and can cause ankylosis and arthritis in both axial and peripheral joints. Although there are many studies showing these limitations nowadays, there is a need to show these limitations with more objective data with the new technology. Evaluating aerobic physical capacity; Cardiopulmonary Exercise Test (KPET) is frequently used in physical performance analysis today. In this study, the investigators want to observe the physical performance differences between 42 AS patients and 42 control group participants by applying KPET and present the expected performance losses in AS patients in the literature with objective data.

DETAILED DESCRIPTION:
AS is an inflammatory disease of unknown etiology, characterized by marked inflammation in the spinal joints and adjacent structures, leading to progressive and ascending bone fusion in the spine. Although peripheral joint involvement is less, hip and shoulder joints are kept in 1/3 of the cases. Inflammatory lesions can also be seen in extraarticular organs such as eyes and heart. Due to joint involvement, limitations in lung capacity, and other extra-articular involvements, physical performance may decrease in AS patients. Both spinal and peripheral joint involvements and pain caused by chronic inflammatory process can lead patients to a more sedentary lifestyle. Therefore, evaluation of physical performance is important in patients with AS. Although there are some methods based on classical observation in evaluating physical performance, Cardiopulmonary Exercise Test (KPET), where objective data about aerobic capacity can be obtained, has been used frequently in scientific studies in recent years. The data such as oxygen consumption, cardiac parameters and speed of the patient on the treadmill in KPET are analyzed numerically; objective performance values such as maximum oxygen use (VO2max), maximum heart rate, and maximum rate can be achieved. It is possible to evaluate all the individuals to whom these tests are applied according to the normal value ranges in the world more clearly in terms of their physical performance and to reshape the exercise program especially according to the missing parameter. For this reason, these methods are preferred primarily in physical performance evaluation in centers with sufficient facilities.

In the literature, although subjective tests and data on physical performance decrease, studies showing clear numerical data are needed. Therefore, in our study; We aim to evaluate the physical performance of patients by applying KPET in our patients with AS diagnosis. Thus, investigators aim to reveal the physical exercise capacity that may be decreased in this patient group with objective numerical data. In addition, patients data will compare with the control group of similar physical characteristics and age.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AS with modified New York Criteria (for AS group)
* Being between the ages of 18-65
* Agree to participate in the study

Exclusion Criteria:

* Cardiac disease
* History of stroke
* Asthma or chronic obstructive pulmonary disease
* Deformity that may prevent exercise
* Hypertension
* Unwilling to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
36-Item Short Form Health Survey (SF-36) | Ten minutes
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The eight sections are:
  vitality,physical functioning,bodily pain,general health perceptions,physical role,functioning,emotional role functioning,social role functioning and mental health.
Bath Ankylosing Spondylitis Disease Activation Index (BASDAI) | Ten minutes
  The BASDAI or Bath Ankylosing Spondylitis Disease Activity Index is a validated diagnostic test which allows a physician, usually a rheumatologist, to determine the effectiveness of a current drug therapy, or the need to institute a new drug therapy for the treatment of Ankylosing spondylitis (AS).The BASDAI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem) in response to six questions asked of the patient pertaining to the five major symptoms of AS:Fatigue, Spinal pain, Arthralgia (joint pain) or swelling, Enthesitis,Morning stiffness duration, Morning stiffness severity
Maximum Oxygen use (VO2max) | 60 minutes
  VO2 max is the maximum rate of oxygen consumption measured during incremental exercise; that is, exercise of increasing intensity.
  The measurement of VO2 max in the laboratory provides a quantitative value of endurance fitness for comparison of individual training effects and between people in endurance training. Maximal oxygen consumption reflects cardiorespiratory fitness and endurance capacity in exercise performance. VO2 max refers to the amount of oxygen a person uses during intense or maximal exercise. Its measurement gives the amount of oxygen consumed per minute for a kilogram of body weight in milliliters.
Maximum heart rate | One minutes
  It is determined by measuring the maximum number of heartbeats observed per minute reached during the KPET.
Maximum speed | One minutes
  It is determined by measuring the maximum average distance traveled per minute on the treadmill in meters / minute.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bezmialem Vakif university, Istanbul
  - BezmialemVU, Istanbul

IPD SHARING:
Plan to Share IPD: No